CLINICAL TRIAL: NCT07075705
Title: Investigating the Feasibility of Using Transperineal Micro-Ultrasound to Detect Clinically Significant Prostate Cancer
Brief Title: Transperineal Micro-ultrasound for the Detection of Prostate Cancer During Biopsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I-4290824; NCI-2025-04490 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-4290824 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2025-07-09; First posted 2025-07-20 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Diagnostic (transperineal micro-ultrasound) (Experimental): Patients undergo transperineal micro-ultrasound imaging over 3 minutes followed by transrectal micro-ultrasound imaging during standard of care prostate biopsy. Patients also undergo MRI during screening.
  Interventions: Procedure: Biopsy of Prostate; Procedure: Magnetic Resonance Imaging; Procedure: Micro-ultrasound Imaging

INTERVENTIONS:
Procedure: Biopsy of Prostate — Undergo standard of care prostate biopsy
  Other Names: Prostate Biopsy; Prostatic Biopsy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Micro-ultrasound Imaging — Undergo transperineal micro-ultrasound imaging
  Other Names: Micro ultrasound; Micro ultrasound Imaging; Micro-ultrasound; microUS
Procedure: Micro-ultrasound Imaging — Undergo transrectal micro-ultrasound imaging
  Other Names: Micro ultrasound; Micro ultrasound Imaging; Micro-ultrasound; microUS

SUMMARY:
This clinical trial studies whether transperineal micro-ultrasound can be used to detect prostate cancer during biopsy. Transrectal ultrasound is often used during prostate biopsy. Transrectal ultrasound imaging is a procedure in which a probe that sends out high-energy sound waves is inserted into the rectum. The sound waves are bounced off internal tissues or organs and make echoes. The echoes form a picture of body tissue called a sonogram. Transrectal ultrasound is used to look for abnormalities in the rectum and nearby structures, including the prostate. The images are used to guide the prostate biopsy. Transperineal micro-ultrasound is completed by placing a probe over the skin between the scrotum and anus (perineum). It is a high-resolution ultrasound at 29 megahertz (MHz) (compared to traditional ultrasound at 6-9 MHz). This higher frequency allows for an improved spatial resolution. This improved spatial resolution is approximately the diameter of a prostatic duct, and therefore, may be able to visualize slight changes in the structure of prostatic ducts that are not possible with standard transrectal ultrasound. Transperineal micro-ultrasound may be more effective in detecting prostate cancer during biopsy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate the feasibility and validity of using transperineal micro-ultrasound to image the prostate and detect clinically significant prostate cancer.

II. To test the quality of visualization of the prostate gland using micro-ultrasound via the transperineal approach.

SECONDARY OBJECTIVE:

I. To compare micro-ultrasound images done via the transperineal method to micro-ultrasound images done via the transrectal method to see if transperineal ultrasound has similar ability to detect suspicious prostate lesions as transrectal micro-ultrasound.

OUTLINE:

Patients undergo transperineal micro-ultrasound imaging over 3 minutes followed by transrectal micro-ultrasound imaging during standard of care prostate biopsy. Patients also undergo magnetic resonance imaging (MRI) during screening.

ELIGIBILITY:
Inclusion Criteria:

* Men aged ≥ 18 years
* Men scheduled for transrectal ultrasound guided prostate biopsy who have had a prebiopsy MRI. Therefore patients unable to have a prebiopsy MRI who have contraindications to MRI or unwilling to undergo MRI would be excluded
* The participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board-approved written informed consent form before receiving any study-related procedure

Exclusion Criteria:

* Any condition which in the investigator's opinion deems the participant an unsuitable candidate for study participation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with Prostate Risk Identification Using Micro-Ultrasound (PRIMUS) score (Feasibility) | Up to 2 months
  At the first stage, 28 patients will be enrolled. If the procedure was successful in at least 18 patients, the procedure will be considered feasible, and the study will proceed to the next stage. If less than 18 successes were observed, the study team will determine whether to continue the trial based on the data collected.
Visualization of the prostate from base to apex with adequate image quality for PRIMUS scoring | Up to 2 months
  Will decide yes or no for whether the prostate can be assessed using transperineal micro ultrasound in order to evaluate for possible prostate cancer using the PRIMUS scoring system. This includes being able to visualize the prostate from base to apex with adequate image quality for PRIMUS scoring.
Visualization of the prostate from right and left lateral margins with adequate image quality for PRIMUS scoring | Up to 2 months
  Will decide yes or no for whether the prostate can be assessed using transperineal micro ultrasound in order to evaluate for possible prostate cancer using the PRIMUS scoring system. This includes being able to visualize the prostate from right and left lateral margins with adequate image quality for PRIMUS scoring.

SECONDARY OUTCOMES:
Successful generation of PRIMUS score in transperineal and transrectal ultrasound images | Up to 7 months
  Will compare transrectal and transperineal micro-ultrasound assessment of PRIMUS score. This will be a yes/no comparison. Summary statistics in frequencies and relative frequencies will be provided.
Ability to visualize the whole prostate using transperineal micro-ultrasound | Up to 7 months
  This will be a yes/no comparison. Summary statistics in frequencies and relative frequencies will be provided.
Quality of images of transperineal ultrasound and transrectal ultrasound of the prostate | Up to 7 months
  The quality of images of transperineal ultrasound will be compared to transrectal ultrasound of the prostate. Summary statistics in frequencies and relative frequencies will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Khurshid A Guru, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States